CLINICAL TRIAL: NCT00472030
Title: An Open Label Case Series on the Effects of Xolair (Omalizumab) in Bullous Pemphigoid
Brief Title: Efficacy and Safety of Omalizumab in Bullous Pemphigoid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Janet Fairley, Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100569
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Results first posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-09

CONDITIONS: Bullous Pemphigoid
Keywords: bullous pemphigoid; omalizumab; xolair; IgE; autoimmunity; skin disease
MeSH Terms: conditions — Pemphigoid, Bullous; Autoimmune Diseases; Skin Diseases | interventions — Omalizumab; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omalizumab (Experimental): Patients will be treated with 150-375 milligrams of Omalizumab (Xolair), based on their baseline weight and serum Immunoglobulin E levels. Omalizumab will be administered subcutaneously on Day 1, and on Week 2, 4, 6, 8, 10, 12 and 14 treatment.
  Interventions: Drug: Omalizumab
- Prednisone (Active Comparator): The control arm of the study will receive standard prednisone therapy to a maximum dose of 0.5 mg/kg/day.
  Interventions: Drug: prednisone

INTERVENTIONS:
Drug: Omalizumab — Patients will be treated with 150-375 milligrams of Omalizumab (Xolair), based on their baseline weight and serum Immunoglobulin E levels. Omalizumab will be administered subcutaneously on Day 1, and on Week 2, 4, 6, 8, 10, 12 and 14 treatment.
  Other Names: Xolair
  Arms: Omalizumab
Drug: prednisone — Prednisone, to a maximum dose of 0.5 mg/kg/day.
  Arms: Prednisone

SUMMARY:
The primary objective is to test the safety and efficacy of Xolair in the treatment of the autoimmune blistering disease, bullous pemphigoid (BP).

This is a pilot, open label case-control study. Patients treated with Xolair will be compared to patients receiving standard treatment with prednisone.

The enrollment period for the study is 24 weeks: 16 weeks active treatment and 8 additional weeks of observation.

DETAILED DESCRIPTION:
Objectives: The primary objective is to test the safety and efficacy of Omalizumab (Xolair) in the treatment of the autoimmune blistering disease, bullous pemphigoid (BP).

Study Rationale: The current treatment for bullous pemphigoid is non-specific immunosuppression, causing great morbidity in these patients. Recently, pathogenic Immunoglogulin Class E autoantibodies have been identified in these patients. Development of a more targeted approach to treatment may reduce morbidity.

Methodology: This is a pilot, open-label case-control study. Patients treated with Omalizumab (Xolair) will be compared to patients receiving standard treatment with prednisone.

Number of centers and patients: This is a single center study that will enroll 12 patients.

Population: Bullous pemphigoid patients, meeting clinical, histological and immunologic criteria for the disease will be enrolled. Pregnant women, children less than 18 years of age, and patients unable to give consent will be excluded from this preliminary study.

Investigational drug: Xolair® (Omalizumab)

Study duration: 24 weeks: 16 weeks of active treatment, 8 additional weeks of observation

Evaluation criteria: Primary: 1. Time to cessation of new blister formation. 2. Percent body surface area of skin involved before and after treatment 3. Total and average daily dose of prednisone required in 30, 60 and 180 days after starting Xolair. Secondary: 1. Number of circulating eosinophils 2. Measurement of circulating anti-BMZ (basement membrane zone) autoantibodies 3. Histamine release assay.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the clinical and histological findings consistent with bullous pemphigoid. Clinically this is defined as urticarial plaques and/or vesicles and bullae. Histologically patients must show characteristic eosinophilic spongiosis and/or subepidermal separation of the skin consistent with BP.
* Patients must have either a positive direct (IgG and/or C3 at the BMZ) or indirect (IgG on the roof of salt-split skin) immunofluorescence microscopy features of pemphigoid.
* Patients of both sexes, all races and ethnic backgrounds that are 18 years of age or older will be eligible to participate in this study.
* Patients much have more than 5% total body surface involved, since patients with less extensive disease are often treated with topical measures only.

Exclusion Criteria:

* Women of childbearing potential not using the contraception method(s) specified during this study. Women of childbearing potential must use proven birth control methods (such as - abstinence, birth control pills, intrauterine device, barrier method combined with gel or foam with spermicide, tubal ligation, or a partner who has had a vasectomy).
* Women who are pregnant or breastfeeding.
* Patients under the age of 18.
* Patients unable to give informed consent.
* Known sensitivity to study drug(s) or class of study drug(s).
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study.
* Any cancer other than non-melanoma skin cancer in the past 5 years.
* All non-melanoma skin cancers must have been adequately treated at entrance to the study.
* Use of any other investigational agent in the last 30 days.
* Treatment with prednisone in the past 2 weeks.
* Weight or serum IgE levels that place the patient outside standard dosing guidelines for Xolair.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet A Fairley, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Department of Dermatology, Iowa City, Iowa, United States

REFERENCES:
- [Background] Dimson OG, Giudice GJ, Fu CL, Van den Bergh F, Warren SJ, Janson MM, Fairley JA. Identification of a potential effector function for IgE autoantibodies in the organ-specific autoimmune disease bullous pemphigoid. J Invest Dermatol. 2003 May;120(5):784-8. doi: 10.1046/j.1523-1747.2003.12146.x. PMID 12713582
- [Background] Fairley JA, Fu CL, Giudice GJ. Mapping the binding sites of anti-BP180 immunoglobulin E autoantibodies in bullous pemphigoid. J Invest Dermatol. 2005 Sep;125(3):467-72. doi: 10.1111/j.0022-202X.2005.23853.x. PMID 16117787
- [Background] Holgate ST, Djukanovic R, Casale T, Bousquet J. Anti-immunoglobulin E treatment with omalizumab in allergic diseases: an update on anti-inflammatory activity and clinical efficacy. Clin Exp Allergy. 2005 Apr;35(4):408-16. doi: 10.1111/j.1365-2222.2005.02191.x. PMID 15836747

RESULTS

PARTICIPANT FLOW:
Groups:
- Omalizumab Treatment Arm: Patients with bullous pemphigoid will be treated with omalizumab for a total treatment period of 14 weeks.
- Prednisone Standard Therapy Treatment Arm: The control arm of the study will receive standard prednisone therapy to a maximum dose of 0.5 milligrams per kilogram per day (mg/kg/day).
Period: Overall Study
Arm/Group | Omalizumab Treatment Arm | Prednisone Standard Therapy Treatment Arm
Started | 2 | 0
Completed | 1 | 0
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Omalizumab Treatment Arm: Patients with bullous pemphigoid will be treated with omalizumab for a total treatment period of 16 weeks.
- Prednisone Standard Therapy Treatment Arm: The control arm of the study will receive standard prednisone therapy to a maximum dose of 0.5 mg/kg/day.
- Total: Total of all reporting groups
Arm/Group | Omalizumab Treatment Arm | Prednisone Standard Therapy Treatment Arm | Total
Number analyzed (Participants) | 2 | 0 | 2
Age Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 2 |  | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 78 (0) |  | 78 (0)
Gender [Number; unit: participants]
  Female | 2 |  | 2
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Median Time From First Dose of Omalizumab Treatment to Cessation of New Blisters.
Description: The study subject underwent physical examination and was assessed for cessation of new blister formation via physical examination and photography.
Time Frame: Up to 24 weeks
Population: The population analyzed included one subject who received Omalizumab treatment on Day 1, Week 2,4,6,8,10,12 and 14 and completed assessments through week 24. A second subject enrolled in the study and received one treatment with Omalizumab and was terminated from the study per investigator at Week 4.
Measure: Number; unit: weeks
Groups:
- Omalizumab Treatment Arm: Omalizumab 150-375 milligrams (mg) will be administered subcutaneously at Day 1, Week 2,4,6,8,10,12, and 14.
Arm/Group | Omalizumab Treatment Arm
Number analyzed (Participants) | 1
weeks | 6

2. Secondary Outcome: Decrease in Anti-BP180 IgG (Immunoglobulin G Anti-Bullous Pemphigoid 180 Antibody) Following Treatment With Omalizumab.
Description: Anti-BP180 IgG levels were completed using an Elisa assay. Anti-BP180 IgG levels were obtained prior to baseline and at week 16
Time Frame: Up to 24 weeks
Population: as for outcome 1
Measure: Number; unit: units per milliliter
Arm/Group | Omalizumab Treatment Arm | Prednisone Standard Therapy Treatment Arm
Number analyzed (Participants) | 1 | 0
units per milliliter | 92.06 |

3. Secondary Outcome: Decrease in Eosinophil Levels Following Treatment With Omalizumab.
Description: The subject's eosinophil count measured at baseline was compared to the eosinophil count at week 8. A normal eosinophil count at the University of Iowa Hospital lab is 0-0.4 cells per microliter
Time Frame: Baseline, 24 weeks.
Population: as for outcome 1
Measure: Number; unit: cells/microliter
Groups:
- Omalizumab Treatment Arm: Patients with bullous pemphigoid will be treated with Omalizumab on Day 1, Week 2,4,6,8,10,12 and 14.
Arm/Group | Omalizumab Treatment Arm | Prednisone Standard Therapy Treatment Arm
Number analyzed (Participants) | 1 | 0
cells/microliter | 2.16 |

4. Primary Outcome: Percent Decrease in the Total Body Surface Area Affected By Active Bullous Pemphigoid Skin Disease From Day 0 to Week 24.
Description: Measurement of total body surface area affected by bullous pemphigoid active skin disease(active erosions, blisters, and/or lesions) was measured at Day 0 (prior to treatment with Omalizumab) and at 24 weeks (24 weeks is end of study).
Time Frame: Up to 24 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of active skin disease
Groups:
- Omalizumab Treatment Arm: Research subjects enrolled to the Omalizumab treatment arm will be treated with Omalizumab on Day 1 and at Week 2,4,6,8,10,12,& 14.
Arm/Group | Omalizumab Treatment Arm
Number analyzed (Participants) | 1
percentage of active skin disease | 22.5

5. Primary Outcome: Median Increase in Prednisone Dosage Measured at Week 4, 8 and 24 in Patients Treated With Omalizumab and in Patients Receiving Standard Therapy.
Description: The total dose of prednisone required to control the bullous pemphigoid at week 4, 8 and 24 weeks was to be calculated in both arms of this study.
Time Frame: Week 4, Week 8 and Week 24
Population: Neither subject required treatment with Prednisone. Since we did not enroll any subject in the Prednisone Standard Therapy Treatment Arm we do not have any measurements for this outcome
Arm/Group | Omalizumab Treatment Arm | Prednisone Standard Therapy Treatment Arm
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Decrease in Anti-BP230 Antibody IgG (Anti-bullous Pemphigoid 230 Antibody Immunoglobulin G) At Baseline and Week 16
Time Frame: Up to 24 weeks
Population: as for outcome 1
Measure: Number; unit: units per milliliter
Arm/Group | Omalizumab Treatment Arm | Prednisone Standard Therapy Treatment Arm
Number analyzed (Participants) | 1 | 0
units per milliliter | 62.6 |

7. Secondary Outcome: Change in Histamine Release Assay Following Treatment With Omalizumab.
Description: The histamine release assay measures the release of histamine which occurs upon stimulation of basophilic granulocytes depending upon their sensitivity to an allergen.
Time Frame: Up to 24 weeks
Population: We were unable to complete this assay in our research subjects due to technical difficulties.
Arm/Group | Omalizumab Treatment Arm | Prednisone Standard Therapy Treatment Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a 24 week time period.
Description: Subjects were underwent physical examination and/or had labwork taken at Baseline/Screening, Week 1,2,4,8,12,16, 20 & 24. Subjects were observed for signs of allergic reaction and vital signs were monitored for two hours after each injection of Omalizumab. Subjects were screened for adverse events throughout the 24 week period.
Arm/Group | Omalizumab Treatment Arm | Prednisone Standard Therapy Treatment Arm
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/0
Other Adverse Events (participants affected / at risk) | 1/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omalizumab Treatment Arm (N=2) | Prednisone Standard Therapy Treatment Arm (N=0)
Hospitalization for Congestive Heart Failure Exacerbation (Cardiac disorders) | 1 (1) | 0 (0) — Subject with known history/treatment of Congestive Heart Failure and chronic obstructive pulmonary disease. ON 8/25/2008, subject experienced shortness of breath with hospitalization, deemed not related to study drug.
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Subject hospitalized for cellulitis at an outside hospital. Subject prescribed antibiotics for skin infection but did not take. Subsequent followup visit revealed Pemphigoid in the site Serious adverse event determined not to be related to study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Omalizumab Treatment Arm (N=2) | Prednisone Standard Therapy Treatment Arm (N=0)
Ankle Edema (Skin and subcutaneous tissue disorders) | 1/1 (1) | 0 (0) — Subject presented with ankle edema at baseline. This was rated as mild, not related to study drug, no action was taken or required and this resolved without sequelae.
Pruritis (Skin and subcutaneous tissue disorders) | 1/1 (1) | 0 (0) — Subject experienced pruritis at baseline. This was rated as moderately severe, unrelated to the study drug, was treated with concomitant medications and was continuing at the end of followup.
Staph Aureus Infection (Skin and subcutaneous tissue disorders) | 1/1 (1) | 0 (0) — Subject was diagnosed with staph aureus infection which was cultured from a superficial skin erosion on the back. This was mild, unrelated to study drug, resolved without sequelae and was treated with concomitant medication.
Nasal Stuffiness (General disorders) | 1/1 (1) | 0 (0) — Subject was diagnosed with nasal stuffiness which was rated as mild in severity, was rated unlikely related to the study drug, was not treated and resolved without sequelae.
Cough associated Nasal Drainage (General disorders) | 1/1 (1) | 0 (0) — Subject experienced a cough associated with nasal drainage which was rated as mild in severity, not treated, resolved without sequelae and rated as unlikely to be related to the study drug use.
Staphylococcus infection (Skin and subcutaneous tissue disorders) | 1/1 (1) | 0 (0) — Subject experienced a staphylococcus infection on the skin of the right toe. This was rated as mild in severity, resolved without sequelae, was rated unlikely to be related to study drug and required the use of concomitant medication.

LIMITATIONS AND CAVEATS:
Limitations of this trial include low enrollment of research subjects and the need to withdraw a subject from the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less